CLINICAL TRIAL: NCT04220892
Title: Pilot Study of Pembrolizumab Combined With Pemetrexed or Abemaciclib for the Treatment of Patients With High Grade Glioma
Brief Title: Pilot Study of Pembrolizumab Combined With Pemetrexed or Abemaciclib for High Grade Glioma
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: One of the study drugs will no longer be supplied by manufacturer and the pembrolizumab + abemaciclib study arm is removed due to toxicity seen in other trials.
Sponsor: Jose Carrillo (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Jose Carrillo, Associate Professor, Neurosciences, Saint John's Cancer Institute
Organization: Saint John's Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JWCI-18-0702 (I3Y-US-I011)
Record Dates: First submitted 2019-11-26; First posted 2020-01-07 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: High Grade Glioma
Keywords: Immunotherapy; Pembrolizumab; Pemetrexed; Abemaciclib; Cyclin-dependent kinase 4 (CDK4); Cyclin-dependent kinase 6 (CDK6); Folate antimetabolite
MeSH Terms: conditions — Glioma | interventions — pembrolizumab; Pemetrexed; abemaciclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pembrolizumab plus Pemetrexed (Experimental): Pembrolizumab plus Pemetrexed
  Interventions: Drug: Pembrolizumab; Drug: Pemetrexed
- Pembrolizumab plus Abemaciclib (Experimental): Pembrolizumab plus Abemaciclib
  Interventions: Drug: Pembrolizumab; Drug: Abemaciclib

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg intravenous (IV) every 3 weeks
  Other Names: Keytruda
Drug: Pemetrexed — 900 mg/m^2 IV every 3 weeks. Supportive medications of ibuprofen, folic acid, vitamin B12, and dexamethasone.
  Other Names: Alimta
  Arms: Pembrolizumab plus Pemetrexed
Drug: Abemaciclib — 150 mg twice a day, by mouth.
  Other Names: Verzenio
  Arms: Pembrolizumab plus Abemaciclib

SUMMARY:
The purpose of this study is to evaluate any preliminary evidence of anticancer activity of pembrolizumab combined with either pemetrexed or abemaciclib when used following surgery and before standard therapy with radiation and temozolomide in patients with newly diagnosed high grade glioma.

Additional aims of the study are to:

* Find out the side effects (good and bad) of pembrolizumab combined with pemetrexed or abemaciclib;
* • Evaluate tumor characteristics by collecting brain tumor tissue samples.
* Measure the amount of pembrolizumab, pemetrexed, and/or abemaciclib that gets in the body by collecting blood and cerebrospinal fluid.
* Look at biomarkers (biochemical features that can be used to measure the progress of disease or the effects of a drug) in blood and cerebrospinal fluid if available.

DETAILED DESCRIPTION:
This is a prospective, open-label, multi-arm exploratory study of pembrolizumab in combination with pemetrexed or abemaciclib for the treatment of adult patients with newly diagnosed high grade glioma. Patients having a clinically planned surgical procedure (biopsy or cytoreduction) for a suspected diagnosis of high grade glioma will be approached for participation in this study. Tumor tissue obtained from surgery will be used for histological diagnosis and clinical molecular profiling, and excess tumor tissue may be collected for potential correlative studies. A small sample of blood and cerebrospinal fluid (CSF) for research will also be collected.

Once a diagnosis of high grade glioma is confirmed, the patient will be allocated to either Treatment Arm 1 (pembrolizumab + pemetrexed), or Treatment Arm 2 (pembrolizumab + abemaciclib). Treatment will be started approximately 7-42 days following surgery once the patient has recovered from surgery. Routine clinical evaluations will be performed prior to treatment initiation and throughout treatment as clinically indicated. Radiographic brain imaging will be performed approximately 21-42 after treatment initiation and then routinely for medical management. Tumor response will be assessed according to immunotherapy Response Assessment in Neuro-Oncology (iRANO) Working Group criteria.

Treatment may continue until the patient experiences unacceptable toxicity or clear disease progression. The determination of whether to stop treatment due to disease progression will be based on the investigator's evaluation of the patient's clinical and radiographic condition, taking into consideration the interpretation of localized inflammatory responses that can mimic radiographic features of tumor progress. Patients discontinuing treatment will be directed by their treating physician to either receive a different treatment regimen (e.g., standard radiation therapy with or without chemotherapy) or undergo a clinically-indicated cytoreductive surgery. If another treatment is started, clinical evaluations and response assessments will continue as clinically-indicated and blood and CSF will be collected after the first month, then every three months.

ELIGIBILITY:
Inclusion Criteria for ALL Arms:

1. Participant or their legal representative has the ability to provide informed consent.
2. Participant has the willingness to comply with all study procedures and availability for the duration of the study.
3. Participant is being evaluated for a potential, or known, diagnosis of high grade glioma.

   Note:Participant must have a diagnosis of high grade (WHO Grade III or IV) glioma following brain surgery to proceed with study treatment.
4. Participant is a candidate for brain surgery.
5. Participant is male or female, ≥ 18 years of age.
6. Participant has a Karnofsky Performance Status ≥ 60%.
7. Participant has adequate organ function:

   1. ANC at least 1.5 x 10^9/L or greater.
   2. Platelets at least 100 x 10^9/L or greater.
   3. Hemoglobin at least 8 g/dL or greater.
   4. Total bilirubin 1.5 x upper limit of normal (ULN) or lower.
   5. ALT and AST 3 x ULN or lower.
   6. Serum creatinine 1.5 x ULN or lower.

Additional Inclusion Criteria for Arm 1 only:

1. Participant has the ability to interrupt nonsteroidal anti-inflammatory (NSAIDS) 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of Pemetrexed.
2. Participant has the ability to take folic acid, Vitamin B12, and dexamethasone according to protocol.
3. Creatinine clearance ≥ 45 mL/min (calculated using standard Cockcroft and Gault formula).

Additional Inclusion Criteria for Arm 1 only:

1. Participant is able to swallow oral medications.

Exclusion Criteria for ALL Arms:

1. Participant has received prior anti-cancer treatment for high-grade glioma.
2. Participant has a diagnosis of immunodeficiency or active autoimmune disease.
3. Participant is receiving chronic systemic steroid therapy in dosing exceeding 8 mg daily of dexamethasone equivalent or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug. This is assessed after surgery, prior to starting drug treatment.
4. Participant has received a live vaccine within 28 days prior to the first dose of study agent. Examples of live vaccines include, but are not limited to measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), typhoid vaccine, and intranasal influenza vaccines (e.g., FluMist®).
5. Participant has a severe or uncontrolled medical disorder that would, in the investigator's opinion, impair ability to receive study intervention, including, but not limited to:

   1. Uncontrolled diabetes;
   2. Renal disease that requires dialysis;
   3. Pulmonary disorder requiring supplemental oxygen to keep saturation >95% and the situation is not expected to resolve within 2 weeks;
   4. Severe dyspnea at rest or requiring oxygen therapy;
   5. Interstitial lung disease;
   6. History of major surgical resection involving the stomach or small bowel;
   7. Preexisting Crohn's disease;
   8. Ulcerative colitis;
   9. Uncontrolled vasculitis and/or disease with known vasculitis;
   10. Preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea;
   11. Psychiatric illness/social situations that would limit compliance with study requirements.
6. Participant has an active bacterial infection requiring intravenous antibiotics at time of initiating study treatment, fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C).
7. Participant has a personal history or presence of any of the following cardiovascular conditions:

   1. Syncope of cardiovascular etiology;
   2. Ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation);
   3. Myocardial infraction within 6 months of investigational product administration;
   4. Unstable angina;
   5. Sudden cardiac arrest;
   6. Congestive heart failure (New York Heart Association classification ≥ 3).
8. Participant is a female of childbearing potential who is pregnant or nursing.

Additional Exclusion Criteria for Arm 1 only:

1. Participant has third space fluid which cannot be controlled by drainage. For patients who develop or have baseline clinically significant pleural or peritoneal effusions (on the basis of symptoms or clinical examination) before or during initiation of pemetrexed therapy, consideration should be given to draining the effusion prior to dosing. However, if, in the investigator's opinion, the effusion represents progression of disease, the patient should be discontinued from study therapy.
2. Transaminases greater than 3.0 x ULN, except in presence of known hepatic metastasis, wherein may be up to 5 x ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-08 (Estimated); Primary Completion 2020-07-08 (Estimated); Study Completion 2020-07-08 (Estimated)

PRIMARY OUTCOMES:
Tumor response rates | one year
  Evidence of anti-tumor activity as measured according to immunotherapy Response Assessment in Neuro-Oncology (iRANO) criteria.

SECONDARY OUTCOMES:
Toxicity assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 4.03. | one year
  Proportion of patients experiencing adverse events
Progression free survival (PFS) | one year
  The duration of time from start of treatment until objective tumor progression or death.
Overall survival (OS) | four years
  The duration of time from start of treatment to death.
Levels of immunotherapeutic agents in specimens | approximately 3 months
  Immunotherapeutic drug levels in specimens.
Change in gene signature of tumor tissue after treatment | approximately 6 months to 2 years
  Comparison of genetic analysis of tumor tissue collected before and after study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Carrillo, MD, Principal Investigator — Saint John's Cancer Institute
Locations (1):
- John Wayne Cancer Institute, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No